CLINICAL TRIAL: NCT03194737
Title: Prostatic Urethral Lift in Subject With Acute Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00004
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-05

CONDITIONS: Acute Urinary Retention; Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH; Urinary retention; prostate; hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention; Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- UroLift System procedure (Experimental): All eligible,enroled subjects will undergo a UroLift procedure.
  Interventions: Device: UroLift System Procedure
- Retrospective Arm (No Intervention): Chart review will be performed on all invasive BPH surgeries (TURP, Holmium Laser Enucleation of the prostate (HoLEP), etc) performed by the site from June 1, 2015 to December 31, 2015

INTERVENTIONS:
Device: UroLift System Procedure — Minimally invasive procedure in patients with acute urinary retention secondary to BPH.
  Other Names: Prostatic UroLift (PUL)
  Arms: UroLift System procedure

SUMMARY:
Assess feasibility and safety of the Prostatic Urethra Lift (PUL) procedure in patients with acute urinary retention secondary to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
The study is a multi-centre, prospective evaluation of PUL and retrospective review of invasive surgery as potential comparator. The study is intended to be conducted at up to 5 different centres in the United Kingdom to enrol up to 50 subjects. Subject follow-up visits are at post-procedure, 6 weeks, 3 months, 6 months and 12 months.

ELIGIBILITY:
UroLift System Procedure Arm

Inclusion Criteria:

1. Male gender
2. Diagnosis of symptomatic BPH
3. Age ≥ 50 years
4. Prostate volume ≤ 100 cc per ultrasound (US)
5. Acute urinary retention with at least one failed trial without catheter (TWOC) while on alpha blocker

Exclusion Criteria:

1. An obstructive or protruding median lobe of the prostate
2. Previous BPH surgical procedure
3. Previous pelvic surgery
4. Urethral conditions that prevents insertion and delivery of device system into bladder
5. Retention volume of >1500 mL
6. Has not had prostate cancer excluded
7. History of prostate or bladder cancer
8. Biopsy of the prostate within the 6 weeks prior to Index Procedure
9. History of neurogenic or atonic bladder
10. Acute or chronic renal failure
11. Known coagulopathies or subject on anticoagulants within 3 days of index procedure (excluding up to 100mg ASA)
12. Known bladder stones within the prior 3 months or treatment within 12 months
13. Prostatitis requiring treatment (antibiotics) within the last year
14. Other co-morbidities that could impact the study results

    * severe cardiac arrhythmias uncontrolled by medications or pacemaker
    * congestive heart failure New York Heart Association (NYHA) III or IV
    * history of uncontrolled diabetes mellitus
    * significant respiratory disease in which hospitalisation may be required
    * known immunosuppression (i.e. AIDS, post-transplant, undergoing chemotherapy)
15. Life expectancy estimated to be less than 5 years
16. Desire to maintain fertility post procedure
17. Unable or unwilling to complete all required questionnaires and follow up assessments
18. Unable or unwilling to sign informed consent form
19. Currently enroled in any other clinical research trial that has not completed the primary endpoint

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Barber, Principal Investigator — Frimley Park Hospital; Oliver Kayes, Principal Investigator — St James's University Hosptial; Mark Rochester, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK); Toby Page, Principal Investigator — Freeman Health System; Rajesh Kavia, Principal Investigator — Central Middlesex Hospital; Nikesh Thiruchelvam, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Freeman Hospital, High Heaton, Newcastle Upon Tyne
  - Frimley Park Hospital, Frimley, Surrey
  - Addenbrooke's Hospital, Cambridge
  - St. James's University Hospital, Leeds
  - Central Middlesex Hospital, London
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Retrospective cohort enrollment was separate from the 52 enrolled in the prospective cohort. Retrospective enrollment was based on a retrospective chart review between Jun 1, 2015 and December 31, 2015.
Period: Overall Study
Arm/Group | UroLift System Procedure | Retrospective Arm
Started | 52 | 49
Completed | 47 | 49
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UroLift System Procedure | Retrospective Arm | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (7.9) | 72.7 (8.0) | 72.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 49 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52 | 49 | 101
Duration of Lower Urinary Tract Symptoms (LUTS) [Count of Participants; unit: Participants]
  <1 year | 12 | 18 | 30
  1-5 years | 19 | 22 | 41
  6-10 years | 12 | 3 | 15
  >=10 years | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Successful Trial Without Catheter Peri-procedurally
Description: Success is defined as a spontaneous voided volume of ≥100 mL associated with a post void residual volume by ultrasound <300 mL 3 days (± 1 day) after the index procedure catheter placement without the need for re-catheterisation.
Time Frame: 3 days (± 1 day) from index procedure
Population: Trial Without Catheter information for retrospective arm was recorded as available from medical record, information from the UroLift System was prospectively collected
Measure: Count of Participants; unit: Participants
Groups:
- UroLift System Procedure: All eligible, enrolled subjects will undergo a UroLift procedure.
  UroLift System Procedure: Minimally invasive procedure in patients with acute urinary retention secondary to BPH.
Arm/Group | UroLift System Procedure | Retrospective Arm
Number analyzed (Participants) | 52 | 49
Participants | 29 | 0

2. Secondary Outcome: Number of Participants With Serious Adverse Events Related to Benign Prostatic Hyperplasia (BPH) Intervention
Description: Number of patients who experienced adjudicated Serious Adverse Events related to Benign prostatic hyperplasia (BPH) Intervention Procedure or Device
Time Frame: Through 3 months
Population: Retrospective arm events were recorded from medical record and was not prospectively collected by sites compared to events collected prospectively from the UroLift System
Measure: Count of Participants; unit: Participants
Arm/Group | UroLift System Procedure | Retrospective Arm
Number analyzed (Participants) | 52 | 49
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Index procedure and up to 1 year
Description: An AE is defined as any undesirable medical occurrence in a clinical trial subject, whether it is considered to be related to the device or not, that includes a clinical sign, symptom, or condition An (SAE) is defined as untoward occurrence that:(a) death; (b) life-threatening; (c) requires hospitalisation or prolongation of existing hospitalisation (d) results in persistent or significant disability or incapacity; or (e) is otherwise considered medically significant by the investigator
Arm/Group | UroLift System Procedure | Retrospective Arm
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 7/52 | 2/49
Other Adverse Events (participants affected / at risk) | 36/52 | 29/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System Procedure (N=52) | Retrospective Arm (N=49)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Blood clot in urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Intestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lucunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System Procedure (N=52) | Retrospective Arm (N=49)
Urinary frequency (Pollakiuria) (Renal and urinary disorders) | 1 (1) | 4 (4)
Dysuria (Renal and urinary disorders) | 9 (9) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Catheter site pain (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Haematuria (Renal and urinary disorders) | 6 (6) | 11 (11)
Incontinence urge (Renal and urinary disorders) | 5 (5) | 2 (2)
Pelvic Pain (Renal and urinary disorders) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 9 (13) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 4 (4)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 8 (8)

LIMITATIONS AND CAVEATS:
Data Retrospectively collected from the invasive Benign prostatic hyperplasia (BPH) surgeries (TURP, Holmium Laser Enucleation of the prostate (HoLEP), etc) was not directly comparable to the prospective UroLIFT system outcomes because of inherent standard of care differences between interventions, standard of care at sites and recording in medical records

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agreements restrict data disclosure until written agreement by or publication by Sponsor

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03194737/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03194737/ICF_001.pdf